CLINICAL TRIAL: NCT00219908
Title: Evaluation of a New Therapeutic Strategy in Early and Active Relapsing-Remitting Multiple Sclerosis: Induction Treatment With Mitoxantrone Followed by Long-Term Treatment With Interferon-beta1b
Brief Title: Evaluation of a New Therapeutic Strategy in Early and Active Relapsing-Remitting Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Bayer (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Farmades, Italy (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 981166
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2005-12-22 (Estimated); Status verified 2005-09

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple sclerosis; Mitoxantrone; Methylprednisolone; Interferon beta1b; Relapse; MRI; EDSS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Recurrence | interventions — Mitoxantrone

INTERVENTIONS:
Drug: Mitoxantrone

SUMMARY:
The aim of the study is to determine whether a therapeutic strategy combining mitoxantrone and interferon beta1b can delay disease progression of at least one point on EDSS scale in patients with clinically very active relapsing-remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* age : 18-45 years,
* Clinical disease satisfying the Poser criteria (Amdmt n°4)
* relapsing-remitting disease (Amdmt N°4)
* at least 2 exacerbations within the preceding 12 months, having left sequelae,
* MRI activity at inclusion expressed by at least one gadolinium-enhanced lesion (cranial MRI with 0.1mmol/kg gadolinium),
* a significant disability at inclusion: EDSS score between 2.5 and 5.5 (Amdt N° 4)
* written informed consent

Exclusion Criteria:

* pregnancy and breast-feeding
* use of an insufficiency effective contraceptive method,
* general immunosuppressive therapy using cyclophosphamide, mitoxantrone,or total lymphoid irradiation
* treatment with azathioprine during the 3 months preceding the study
* clinical relapse or intensive corticosteroid treatment within the 30 days preceding inclusion,
* associated disease (psychiatric disorder, depressive statenot controlled by appropriate drug therapy, history of heart disease at inclusion examination

Ages: 18 Years to 45 Years | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124
Dates: Start 1999-07; Study Completion 2006-06

PRIMARY OUTCOMES:
Time to confirmed progression of at least one EDSS point during the 3 years of the study.

SECONDARY OUTCOMES:
- percentage of patients with confirmed progression of at least one point EDSS (confirmed at 3 and 6 months) during the 3 years of the study,
- annual rate of relapse;
- percentage of relapse-free patients during the study period,
- quality of life,
- percentage of patients without evidence of disease activity on serial MRIs at months 9, 24 and 36 (number of contrast-enhanced lesions on the annual MRIs, change in lesion burden).

CONTACTS AND LOCATIONS:
Overall Officials: Gilles EDAN, Professor, Study Director — CHU Rennes
Locations (23):
- France (17):
  - Hôpital Cote de Nacre, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - Hôpital Général, Dijon
  - CHU Limoges, Limoges
  - Institut Catholique de Lille, Lomme
  - Pierre Weitheimer Hospital, Lyon
  - Chu Timone, Marseille
  - Centre Guy de Chauliac, Montpellier
  - CHU Hôpital Central, Nancy
  - CHU, Nice
  - CHU Pitié-Salpétrière, Paris
  - Hôpital Saint-Anne, Paris
  - Centre Fondation Rotschild, Paris
  - Tenon Hospital, Paris
  - CHU Strasbourg, Strasbourg
  - CHU Purpan, Toulouse
- Italy (6):
  - Psichiatriche dell'Università di Bari, Policlinico, Bari
  - Dipartimento di Scienze Neurologiche e Psichiatriche, Florence
  - Hospedal Civile, Gallarate
  - Neuroriabilitazione dell'Università, Genova
  - Fondazionz SAN Raffaele del monte tabor, Milan
  - Clinica Neurologica Università di Torino, Torino